CLINICAL TRIAL: NCT03263897
Title: Feasibility of Using a Mobile Device Controlled Micro-pressure Pulse Insufflator for Acute Migraine Relief
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Manufacturer's decision
Sponsor: Caps Research Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CI-IRB-20170814001
Record Dates: First submitted 2017-08-23; First posted 2017-08-28 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Migraine
Keywords: abortive effect; mobile interface
MeSH Terms: conditions — Migraine Disorders | interventions — Insufflation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active (Experimental): Receiving insufflation during an acute episode of migraine in both visits
  Interventions: Device: insufflation
- Sham (Sham Comparator): Receiving placebo insufflation during an acute episode of migraine in the first visit and receiving insufflation during an acute episode in the second visit
  Interventions: Device: insufflation; Device: placebo insufflation

INTERVENTIONS:
Device: insufflation — mobile interface driven insufflation of the ear canal
Device: placebo insufflation — mobile interface driven placebo insufflation of the ear canal
  Arms: Sham

SUMMARY:
Evaluate the feasibility of using a mobile interface to control the insufflator device administering treatment for aborting (stopping) an acute episode of migraine. The patient, under clinical supervision, will use the mobile interface to "self administer" the treatment when experiencing an acute episode of migraine. The supervising clinician will monitor the patient and the device to make sure that no harm could come to the patient and will be ready to intervene if any adverse effects were suspected to or in the process of happening.

DETAILED DESCRIPTION:
After signing the consent form and being enrolled in the study, the subject will be asked to answer an enrollment questionnaire on the general characteristics of the migraine attacks he or she is suffering. Then, the subject will be instructed to call 1-800 number to notify the clinic that they have a migraine.

Upon presentation with an acute migraine attack, the patient will be randomly assigned to two groups: an active comparator and a sham comparator. During the first session, the active group will receive the actual treatment whereas the placebo group will receive a sham treatment (using an exact replica of the device with the same software and hardware controls that delivers a simulated treatment with no actual pressure delivered - only a simulation of mechanical functions and sounds to simulate an actual treatment). During the second treatment, both groups will receive the actual treatment.

During either session, upon presentation with an acute migraine attack, the subject will be assessed by taking blood pressure, pulse, temperature, subjective pain score on a scale of 0-10 (similar to the scales used in the device's interface) and on a scale from 0 to 3 (typically used in headache studies to establish the pain level) as well as subjective associated symptoms scores on the same 0-10 scale. Bilateral otoscopic examination will be used to confirm intact tympanic membranes to ensure that subjects can safely receive the treatment. Also, subjects will receive bilateral hearing screening and their ability to maintain balance will be assessed. Then the subjects will be attached to a comfortable heart rate variability (HRV) monitor and asked to lie down quietly for 5 min so as to obtain a baseline HRV recording. Soft silicone ear plugs will be inserted in the subject's ears. These plugs are attached to the automated insufflator device (active or sham, depending on the group the subject is assigned to). The subject will control the device using a mobile app: an easy to use interface will allow the subject to provide the device all the information needed for the automatic selection of the treatment protocol most appropriate for the subject. Once selected, the treatment will last 30 minutes. The subjects heart rate, HRV, and pulse oxygenation will be monitored throughout the insufflation procedure to measure physiologic response to the procedure as well as to bolster the safety of the procedure. The heart rate and pulse Ox values will be recorded every minute (heart rate and pulse ox) on the vitals form, the HRV will be a continuous recording for the entire duration of the treatment. After 10 and 20min of treatment, the subject will be asked the corresponding pain score on a scale of 0-10. Vitals will be taken again at the end of the treatment. The subject will then be asked to lie again quietly for 5 mins as a final HRV recording is obtained for comparison against the pre-evaluation one. Bilateral hearing and ability to maintain balance will also be screened again at the end of the treatment and compared with the pre-treatment measures to see if they were affected by the treatment.

Subjective pain and symptom scores will be obtained immediately after the 30min treatment, and at the 2 hour post and 24 hour post treatment end points. Each user will receive only a single treatment, administered in the clinic setting. 2 hour and 24 hour end point assessments will be obtained telephonically.

The second visit will follow the identical procedure with the exception that all subjects will receive an actual treatment at this stage.

Independently whether they come back for the second visit, subjects will be questioned by telephone one calendar month after their first treatment as to the number, type and intensity of migraines experienced in the period between the first treatment and the 1-month follow up phone call.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects suffering from acute migraine episodes
* Possibly located in the Phoenix, AZ area

Exclusion Criteria:

* Pregnant/nursing women

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in Symptoms severity scale | Baseline, immediately post-treatment
  Subjects will grade the severity of their symptoms on a scale from 0 to 10. Changes in the symptoms severity scale will be assessed between pre and immediately post treatment
Changes in pain level | Baseline, immediately post-treatment
  Subjects will grade their pain level on a scale from 0 to 10 as well as on another scale from 0 to 3. Changes in the pain level scale will be assessed between pre and immediately post treatment

SECONDARY OUTCOMES:
Changes in Symptoms severity scale at 2 hours | Baseline, 2 hours post-treatment
  Subjects will grade the severity of their symptoms on a scale from 0 to 10. Changes in the symptoms severity scale will be assessed between pre and 2h post treatment
Changes in Symptoms severity scale at 24 hours | Baseline, 24 hours post-treatment
  Subjects will grade the severity of their symptoms on a scale from 0 to 10. Changes in the symptoms severity scale will be assessed between pre and 24h post treatment
Changes in pain level at 2 hours | Baseline, 2 hours post-treatment
  Subjects will grade their pain level on a scale from 0 to 10 as well as on another scale from 0 to 3. Changes in the pain level scale will be assessed between pre and 2h post treatment
Changes in pain level at 24 hours | Baseline, 24 hours post-treatment
  Subjects will grade their pain level on a scale from 0 to 10 as well as on another scale from 0 to 3. Changes in the pain level scale will be assessed between pre and 24h post treatment

CONTACTS AND LOCATIONS:
Overall Officials: David M George, DC, Principal Investigator — GBS Ventures
Locations (2):
- United States (2):
  - YRMC: Physiatry, Neurosurgery, Neurology Clinic, Prescott, Arizona
  - FNOR Clinic Scottsdale, Scottsdale, Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] D.M. George, G. Pagnacco, K.E. Willey, J.P. Claude, E. Oggero "SAFETY AND USABILITY FACTORS IN DEVELOPMENT OF A NOVEL, AUTOMATED TREATMENT DEVICE FOR ACUTE MIGRAINE", Biomedical Sciences Instrumentation, 2017, Vol. 53, pp 398-403.